CLINICAL TRIAL: NCT06858332
Title: Lipoprotein(a) Levels in Patients With Atherosclerotic Cardiovascular Diseases in Russia
Acronym: STaRT
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CTQJ230A1RU01
Record Dates: First submitted 2025-02-18; First posted 2025-03-05 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: lipoprotein(a),; ASCVD,; cardiovascular disease,; CVD
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases | interventions — Atorvastatin; Simvastatin; Ezetimibe; Niacin; ciprofibrate; Fenofibrate; Bezafibrate; evolocumab; alirocumab; ALN-PCS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- ASCVD patients: Patients aged 18 and above with a history of ASCVD including peripheral arterial revascularization
  Interventions: Drug: Atorvastatin; Drug: Simvastatin; Drug: Rozuvastatin; Drug: Ezetimibe; Drug: Niacin; Drug: Ciprofibrate; Drug: Fenofibrate; Drug: Bezafibrate; Drug: Evolocumab; Drug: Alirocumab; Drug: Inclisiran
- Relatives of the ASCVD patients: A first-degree relative of the ASCVD patient (patient's parents and children) with Lp(a) ≥125 nmol/L.
  Interventions: Drug: Atorvastatin; Drug: Simvastatin; Drug: Rozuvastatin; Drug: Ezetimibe; Drug: Niacin; Drug: Ciprofibrate; Drug: Fenofibrate; Drug: Bezafibrate; Drug: Evolocumab; Drug: Alirocumab; Drug: Inclisiran

INTERVENTIONS:
Drug: Atorvastatin — 3-Hydroxy-3-methylglutaryl-CoA reductase inhibitors (statins)
Drug: Simvastatin — 3-Hydroxy-3-methylglutaryl-CoA reductase inhibitors (statins)
Drug: Rozuvastatin — 3-Hydroxy-3-methylglutaryl-CoA reductase inhibitors (statins)
Drug: Ezetimibe — Ezetimibe
Drug: Niacin — Niacin
Drug: Ciprofibrate — Fibrates
Drug: Fenofibrate — Fibrates
Drug: Bezafibrate — Fibrates
Drug: Evolocumab — PCSK9 inhibitor
Drug: Alirocumab — PCSK9 inhibitor
Drug: Inclisiran — Small interfering RNA

SUMMARY:
This study has the purpose to answer how the Lipoprotein(a) (Lp(a)) level is distributed among Atherosclerotic cardiovascular disease (ASCVD) patients in Russia, and what is the connection between elevated levels of this parameter and the cardiovascular disease (CVD) risk.

DETAILED DESCRIPTION:
This study will consist of several phases (consecutive stages):

Phase I: a cross-sectional study of Lp(a) level with ASCVD patients

Phase II:

* A non-interventional, prospective, cohort study with the phase I patients
* A cross-sectional study of Lp(a) levels with relatives of phase I patients
* A non-interventional, prospective, cohort study with patients' relatives

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (signed and dated).
2. Males and females aged ≥18 years.
3. Presence of one of the following ASCVDs for at least 3 months within the 2 years prior to signing the informed consent to participate in this study:

   * history of MI;
   * history of IS and/or TIA;
   * IHD confirmed by coronary angiography (stenosis ≥50%);
   * any revascularization surgery (emergency or planned), including CABG, PCI, carotid endarterectomy or carotid/intracranial stenting;
   * peripheral artery disease (intermittent claudication with ankle-brachial index ≤0.90 and/or lower limb amputation or revascularization in case of lower limb ischemia).

Exclusion Criteria:

1. Acute infectious and inflammatory diseases, such as COVID-19, in the month leading up to the Screening visit.
2. Lp(a)-lowering therapy/methods (Lp(a) apheresis with PCSK9 inhibitors, inclisiran prior to the Screening visit) in the medical history before the Screening visit.
3. Participation in any interventional clinical study with investigational or marketed medicinal products at the time of enrollment.
4. Participation in other real-world clinical studies.
5. Stages 4 and 5 of chronic kidney disease (glomerular filtration rate CKD-EPI <30 mL/min/1.73 m2) and/or hepatic disease (total bilirubin: 2 × ULN).

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the history of atherosclerotic cardiovascular disease (ASCVD). First-degree relatives of the ASCVD patient (patient's parents and children) with Lp(a) ≥125 nmol/L
Sampling Method: Probability Sample
Enrollment: 2382 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients (%) with Lp(a) ≥125 nmol/L | Baseline
  Percentage of patients (%) with Lp(a) ≥125 nmol/L at baseline
The difference in the number of patients with cardiovascular events (%) between the groups | 24 months
  The difference in the number of patients (%) with new cardiovascular events between the groups of patients with elevated Lp(a) ≥125 nmol/L and Lp(a) <125 nmol/L

SECONDARY OUTCOMES:
Percentage of patients (%) with at least one CVD, and ASCVD number in different subgroups stratified by Lp(a) level | Baseline
  Percentage of patients (%) with at least one CVD by Lp(a) level: ≤25 nmol/L, 25-75 nmol/L, 75-125 nmol/L, 125-188 nmol/L, 188-250 nmol/L, ≥250 nmol/L
  *CVD - Cardiovascular disease; ASCVD - Atherosclerotic cardiovascular disease
Percentage of ASCVD patients (%) in accordance with the Lp(a) level | Baseline
  Percentage of ASCVD patients (%) by Lp(a) level: ≤25 nmol/L, 25-75 nmol/L, 75-125 nmol/L, 125-188 nmol/L, 188-250 nmol/L, ≥250 nmol/L
Age of patients at the time of the first ASCVD in different subgroups in accordance with the Lp(a) level | Baseline
  Age of patients at the time of the first ASCVD in different subgroups by Lp(a) level: ≤25 nmol/L, 25-75 nmol/L, 75-125 nmol/L, 125-188 nmol/L, 188-250 nmol/L, ≥250 nmol/L
Percentage of patients (%) with disability groups I, II, and III in different subgroups stratified by the Lp(a) level | Baseline
  Percentage of patients (%) with disability groups I, II, and III in different subgroups stratified by the Lp(a) level: ≤25 nmol/L, 25-75 nmol/L, 75-125 nmol/L, 125-188 nmol/L, 188-250 nmol/L, ≥250 nmol/L
Age of assignment of any disability group in different subgroups by the Lp(a) level | Baseline
  Age of assignment of any disability group in different subgroups by the Lp(a) level: ≤25 nmol/L, 25-75 nmol/L, 75-125 nmol/L, 125-188 nmol/L, 188-250 nmol/L, ≥250 nmol/L
Duration of temporary incapacity (sick leave) following the onset of CVE in different subgroups based on Lp(a) level | Baseline
  Duration of temporary incapacity (sick leave) following the onset of CVE (cardiovascular event) in different subgroups based on Lp(a) level: ≤25 nmol/L, 25-75 nmol/L, 75-125 nmol/L, 125-188 nmol/L, 188-250 nmol/L, ≥250 nmol/L
Percentage of patients (%) without an official disability status who had to completely stop working after developing CVE in different subgroups based on Lp(a) level | Baseline
  Percentage of patients (%) without an official disability status who had to completely stop working after developing CVE (cardiovascular event) in different subgroups based on Lp(a) level: ≤25 nmol/L, 25-75 nmol/L, 75-125 nmol/L, 125-188 nmol/L, 188-250 nmol/L, ≥250 nmol/L
Lp(a) distribution level by a ASCVD type | Baseline
  Percentage of patients with peripheral artery disease (PAD), ischemic stroke (IS), ischemic heart disease by the Lp(a) level*
  *≤25 nmol/L, 25-75 nmol/L, 75-125 nmol/L, 125-188 nmol/L, 188-250 nmol/L, ≥250 nmol/L
Percentage (%) of ASCVD patients with elevated Lp(a) levels by gender and age (20-30, 31-40, 41-50, 51-60, 61-70, 71-80, 81-90 years) | Baseline
  Percentage (%) of ASCVD patients with elevated Lp(a) levels by gender and age (20-30, 31-40, 41-50, 51-60, 61-70, 71-80, 81-90 years)
Percentage of patients (%) with hemodynamically significant coronary atherosclerosis (stenosis ≥50%) in different subgroups by the Lp(a) level | Baseline
  Percentage of patients (%) with hemodynamically significant coronary atherosclerosis (stenosis ≥50%) in different subgroups by the Lp(a) level ≤25 nmol/L, 25-75 nmol/L, 75-125 nmol/L, 125-188 nmol/L, 188-250 nmol/L, ≥250 nmol/L
Percentage of ASCVD patients (%) with elevated Lp(a) levels in groups stratified by the number of coronary arteries with hemodynamically significant stenosis in patients with relevant available data | Baseline
  Percentage of ASCVD patients (%) with elevated Lp(a) levels in groups stratified by the number of coronary arteries with hemodynamically significant stenosis in patients with relevant available data
Percentage (%) of ASCVD patients with an elevated Lp(a) level classified depending on the presence of multifocal atherosclerosis, ischemic heart disease, and peripheral artery disease | Baseline
  Percentage (%) of ASCVD patients with an elevated Lp(a) level classified depending on the presence of multifocal atherosclerosis, ischemic heart disease, and peripheral artery disease
Percentage of ASCVD patients (%) with elevated Lp(a) levels classified into groups with different numbers of MI events | Baseline
  Percentage of ASCVD patients (%) with elevated Lp(a) levels classified into groups with different numbers of myocardial infarction (MI) events
Percentage of ASCVD patients (%) with elevated Lp(a) levels classified into groups with different numbers of IS and TIA events | Baseline
  Percentage of ASCVD patients (%) with elevated Lp(a) levels classified into groups with different numbers of ischemic stroke (IS) and transient ischemic attack (TIA) events
Percentage of ASCVD patients (%) with elevated Lp(a) levels classified into groups with different types of hospitalization (planned/emergency) | Baseline
  Percentage of ASCVD patients (%) with elevated Lp(a) levels classified into groups with different types of hospitalization (planned/emergency)
Percentage (%) of ASCVD patients with elevated Lp(a) levels classified by the first cardiovascular event (CVE) | Baseline
  Percentage (%) of ASCVD patients with elevated Lp(a) levels classified by the first CVE (any of the following: myocardial infarction, ischemic stroke, transient ischemic attack, percutaneous coronary intervention, etc.)
Percentage of ASCVD patients (%) with elevated Lp(a) levels by the PCI number (planned/emergency) | Baseline
  Percentage of ASCVD patients (%) with elevated Lp(a) levels by the percutaneous coronary intervention (PCI) number (planned/emergency)
Percentage of patients (%) with the first CVE (MI or IS) (before the Screening visit) in different subgroups by the Lp(a) level | Baseline
  Percentage of patients (%) with the first CVE (MI or IS) (before the Screening visit) in different subgroups by the Lp(a) level ≤25 nmol/L, 25-75 nmol/L, 75-125 nmol/L, 125-188 nmol/L, 188-250 nmol/L, ≥250 nmol/L
Percentage of patients (%) with several CVEs (MI or IS) (before the Screening visit) in different subgroups by the Lp(a) level | Baseline
  Percentage of patients (%) with several CVEs (MI or IS) (before the Screening visit) in different subgroups by the Lp(a) level ≤25 nmol/L, 25-75 nmol/L, 75-125 nmol/L, 125-188 nmol/L, 188-250 nmol/L, ≥250 nmol/L
Number of recurrent CVEs in different subgroups by the Lp(a) level | Baseline
  Number of recurrent CVEs in different subgroups by the Lp(a) level ≤25 nmol/L, 25-75 nmol/L, 75-125 nmol/L, 125-188 nmol/L, 188-250 nmol/L, ≥250 nmol/L
Percentage of patients (%) with unstable angina, manifestations of TIA, PCI, and CABG in medical history (before the Screening visit) in different subgroups by the Lp(a) level | Baseline
  Percentage of patients (%) with unstable angina, manifestations of transient ischemic attack (TIA), percutaneous coronary intervention (PCI), and coronary artery bypass grafting (CABG) in medical history (before the Screening visit) in different subgroups by the Lp(a) level ≤25 nmol/L, 25-75 nmol/L, 75-125 nmol/L, 125-188 nmol/L, 188-250 nmol/L, ≥250 nmol/L
Percentage of patients (%) with multiple CVE, such as unstable angina, TIA, PCI, and CABG (before or after the index/screening visit), in different subgroups based on Lp(a) level | Baseline
  Percentage of patients (%) with multiple CVE, such as unstable angina, transient ischemic attack (TIA), percutaneous coronary intervention (PCI), and coronary artery bypass grafting (CABG) (before or after the index/screening visit), in different subgroups based on Lp(a) level ≤25 nmol/L, 25-75 nmol/L, 75-125 nmol/L, 125-188 nmol/L, 188-250 nmol/L, ≥250 nmol/L
Percentage of patients (%) with severe CVE (MI, IS) (after the index/screening visit) based on the Lp(a) level in different subgroups | 3, 9, 12, 18, and 24 months
  Percentage of patients (%) with severe CVE (MI, IS) based on the Lp(a) level ≤25 nmol/L, 25-75 nmol/L, 75-125 nmol/L, 125-188 nmol/L, 188-250 nmol/L, ≥250 nmol/L at 3, 9, 12, 18, and 24 months
Number of patients with recurrent CVEs (more than one event during the follow-up period) and the mean number of recurrent complications in the post-index visit period | 3, 9, 12, 18, and 24 months
  Number of patients with recurrent CVEs (more than one event during the follow-up period) and the mean number of recurrent complications at 3, 9, 12, 18, and 24 months
Percentage of patients (%) with cardiovascular deaths after the index/screening visit in different subgroups by the Lp(a) level | 3, 9, 12, 18, and 24 months
  Percentage of patients (%) with cardiovascular deaths in different subgroups by the Lp(a) level ≤25 nmol/L, 25-75 nmol/L, 75-125 nmol/L, 125-188 nmol/L, 188-250 nmol/L, ≥250 nmol/L at 3, 9, 12, 18, and 24 months
Percentage of patients who died after the index/screening visit in different subgroups by the Lp(a) level | 3, 9, 12, 18, and 24 months
  Percentage of patients who died in different subgroups by the Lp(a) level ≤25 nmol/L, 25-75 nmol/L, 75-125 nmol/L, 125-188 nmol/L, 188-250 nmol/L, ≥250 nmol/L at 3, 9, 12, 18, and 24 months
Percentage of patients (%) who needed emergency medical care or visited a medical facility during the period following the index/screening visit in different subgroups by the Lp(a) level | 3, 9, 12, 18, and 24 months
  Percentage of patients (%) who needed emergency medical care or visited a medical facility in different subgroups by the Lp(a) level ≤25 nmol/L, 25-75 nmol/L, 75-125 nmol/L, 125-188 nmol/L, 188-250 nmol/L, ≥250 nmol/L at 3, 9, 12, 18, and 24 months
Number of emergency visits or visits to a medical facility following the index/screening visit in various subgroups by the Lp(a) level | 3, 9, 12, 18, and 24 months
  Number of emergency visits or visits to a medical facility in various subgroups by the Lp(a) level ≤25 nmol/L, 25-75 nmol/L, 75-125 nmol/L, 125-188 nmol/L, 188-250 nmol/L, ≥250 nmol/L at 3, 9, 12, 18, and 24 months
Percentage of ASCVD patients (%) who achieved the target LDL-C level with the current lipid-lowering therapy | 3, 9, 12, 18, and 24 months
  Percentage of ASCVD patients (%) who achieved the target LDL-C level with the current lipid-lowering therapy
Percentage of ASCVD patients (%) receiving lipid-lowering therapy, who experienced a change in Lp(a) levels | 3, 9, 12, 18, and 24 months
  Percentage of ASCVD patients (%) receiving lipid-lowering therapy, who experienced a change in Lp(a) levels
Number of first-degree relatives (%) of patients with Lp(a) ≥125 nmol/ | Baseline
  Number of first-degree relatives (%) of patients with Lp(a) ≥125 nmol/L
Difference between groups in the number of relatives (%) with CVD complications during the 2-year observation period | 24 months
  The difference in the number of relatives (%) with new cardiovascular events between the groups of patients with elevated Lp(a) ≥125 nmol/L and Lp(a) <125 nmol/L

CONTACTS AND LOCATIONS:
Locations (16):
- Russia (16):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kaluga
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Krasnoyarsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Omsk
  - Novartis Investigative Site, Perm
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Surgut
  - Novartis Investigative Site, Tomsk
  - Novartis Investigative Site, Tyumen
  - Novartis Investigative Site, Vladimir
  - Novartis Investigative Site, Vladivostok
  - Novartis Investigative Site, Voronezh
  - Novartis Investigative Site, Yakutsk
  - Novartis Investigative Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No